CLINICAL TRIAL: NCT02124746
Title: Open-label Study to Assess the Long-term Safety and Efficacy of Momelotinib in Subjects With Primary Myelofibrosis, Post-polycythemia Vera Myelofibrosis, Post Essential Thrombocythemia Myelofibrosis, Polycythemia Vera or Essential Thrombocythemia
Brief Title: Long-term Safety and Efficacy of Momelotinib in Subjects With Primary Myelofibrosis, Post-polycythemia Vera Myelofibrosis, Post-essential Thrombocythemia Myelofibrosis, Polycythemia Vera or Essential Thrombocythemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sierra Oncology LLC - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-352-1154; 2013-004476-36 (EudraCT Number)
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Results first posted 2021-02-05 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Primary Myelofibrosis; Post-Polycythemia Vera Myelofibrosis; Post-Essential Thrombocythemia Myelofibrosis; Polycythemia Vera; Essential Thrombocythemia
Keywords: Primary Myelofibrosis; Post Polycythemia Vera Myelofibrosis; Post Essential Thrombocythemia Myelofibrosis; Polycythemia Vera; Essential Thrombocythemia; blood disorders
MeSH Terms: conditions — Primary Myelofibrosis; Polycythemia Vera; Thrombocythemia, Essential; Hematologic Diseases | interventions — N-(cyanomethyl)-4-(2-((4-(4-morpholinyl)phenyl)amino)-4-pyrimidinyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Participants previously enrolled in Study CCL09191E will receive momelotinib for approximately 4 years.
  Interventions: Drug: Momelotinib
- Cohort 2 (Experimental): Participants previously enrolled in Study YM387-II-02 will receive momelotinib for approximately 4 years.
  Interventions: Drug: Momelotinib
- Cohort 3 (Experimental): Participants previously enrolled in Study GS-US-354-0101 will receive momelotinib for up to 4 years.
  Cohort 3 was closed and all enrolled participants were discontinued from this study because parent Study GS-US-354-0101 was terminated.
  Interventions: Drug: Momelotinib
- Cohort 4 (Experimental): Participants previously enrolled in Study GS-US-352-1672 will receive momelotinib for approximately 4 years.
  Interventions: Drug: Momelotinib

INTERVENTIONS:
Drug: Momelotinib — Momelotinib tablets administered orally once daily
  Other Names: GS-0387; CYT387

SUMMARY:
This open-label study is to determine the long-term safety and tolerability of momelotinib in previously enrolled study participants with primary myelofibrosis (PMF), post-polycythemia vera myelofibrosis (post-PV MF), post-essential thrombocythemia myelofibrosis (post-ET MF), polycythemia vera (PV), or essential thrombocythemia (ET), who have tolerated and achieved stable disease or better with momelotinib treatment while enrolled in a previous clinical trial.

ELIGIBILITY:
Key Inclusion Criteria:

* Currently enrolled in study CCL09101E, or YM387-II-02, or successfully completed 24 weeks of study GS-US-352-1672
* Able to comprehend and willing to sign informed consent form

Key Exclusion Criteria:

* Known hypersensitivity to momelotinib, its metabolites, or formulation excipients

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2014-04-30 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2018-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (22):
- United States (15):
  - Scottsdale, Arizona
  - Orange, California
  - Stanford, California
  - Whittier, California
  - Jacksonville, Florida
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Rochester, Minnesota
  - St Louis, Missouri
  - New York, New York
  - The Bronx, New York
  - Cleveland, Ohio
  - Houston, Texas
  - Salt Lake City, Utah
- Australia (2):
  - Frankston, Victoria
  - Parkville, Victoria
- Canada (2):
  - Toronto, Ontario
  - Montreal, Quebec
- France (2):
  - La Tronche
  - Paris
- Minden, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Benefiting subjects enrolled in 1 of 3 prior momelotinib (MMB) studies (parent studies) for the treatment of MF were included for continued dosing of MMB. Cohort 3 (PV/ET; n=13) was closed and subjects were discontinued due to limited efficacy of MMB in the treatment of PV/ET observed in the parent study. Cohort 3 was excluded from all analyses.
Groups:
- Cohort 1 (CCL09101/ CCL09101E/ GS-US-352-1154): Subjects with PMF, post-PV MF or post-ET MF previously enrolled in parent study CCL09101/ CCL09101E.
- Cohort 2 (YM387-II-02/GS-US-352-1154): Subjects with PMF, post-PV MF or post-ET MF previously enrolled in parent study YM387-II-02.
- Cohort 4 (GS-US-352-1672/GS-US-352-1154): Subjects with PMF, post-PV MF or post-ET MF previously enrolled in parent study GS-US-352-1672.
Period: Overall Study
Arm/Group | Cohort 1 (CCL09101/ CCL09101E/ GS-US-352-1154) | Cohort 2 (YM387-II-02/GS-US-352-1154) | Cohort 4 (GS-US-352-1672/GS-US-352-1154)
Started | 30 | 22 | 22
Completed | 11 | 4 | 0
Not Completed | 19 | 18 | 22
Not completed — Adverse Event | 2 | 1 | 2
Not completed — Death | 2 | 1 | 3
Not completed — Lack of Efficacy | 3 | 2 | 2
Not completed — Physician Decision | 6 | 4 | 5
Not completed — Non-Compliance with Study Drug | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 6
Not completed — Disease Progression | 3 | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (CCL09101/ CCL09101E/ GS-US-352-1154) | Cohort 2 (YM387-II-02/GS-US-352-1154) | Cohort 4 (GS-US-352-1672/GS-US-352-1154) | Total
Number analyzed (Participants) | 30 | 22 | 22 | 74
Age, Continuous [Median (Full Range); unit: years] | 66.0 [34.0 to 82.0] | 64.0 [48.0 to 80.0] | 68.0 [44.0 to 88.0] | 66.5 [34.0 to 88.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 10 | 9 | 36
  Male | 13 | 12 | 13 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 26 | 20 | 18 | 64
  Black or African American | 0 | 2 | 2 | 4
  Asian | 2 | 0 | 0 | 2
  Hispanic or Latino | 1 | 0 | 0 | 1
  Other | 1 | 0 | 2 | 3
Transfusion Dependent (at baseline in parent study) [Count of Participants; unit: Participants]
  Yes | 7 | 7 | 22 | 36
  No | 23 | 12 | 0 | 35
  Missing | 0 | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Long Term Safety and Tolerability as Measured by the Incidence and Severity of Adverse Events and Clinical Laboratory Abnormalities
Description: Long-term safety and tolerability profile of momelotinib based on safety data (adverse events and selected hematology and chemistry laboratory parameters) collected after the first dose of momelotinib in the parent study.
Time Frame: From the first dose of momelotinib in the parent study to 30 days following permanent discontinuation of momelotinib in Study GS-US-352-1154.
Population: It was pre-specified that safety outcomes would be analyzed and summarized by starting dose in Study GS-US-352-1154. Therefore data for this outcome measure are presented for the total subjects enrolled to Study GS-US-352-1154 and not by cohort.
Measure: Count of Participants; unit: Participants
Groups:
- Total: All subjects enrolled to Study GS-US-352-1154
Arm/Group | Total
Number analyzed (Participants) | 74
Participants
  Subjects with ≥ one AE (any grade) | 73
  Subjects with ≥ one Grade 3 or higher AE | 62
  Subjects with Grade 3 lab toxicity (highest grade) | 36
  Subjects with Grade 4 lab toxicity (highest grade) | 16

2. Secondary Outcome: Splenic Response Rate
Description: The number of subjects achieving a spleen response, defined as a reduction of 50% or more in palpable splenomegaly of a spleen that was at least 10 cm below the LCM at baseline, or a spleen that was palpable at > 5 cm and < 10 cm below the LCM at baseline becoming not palpable for at least 56 days, using baseline of the parent study as the reference.
Time Frame: From baseline in the parent study until the last spleen assessment in Study GS-US-352-1154, up to 30 days following permanent discontinuation of momelotinib.
Population: Subjects with splenomegaly >5 cm at baseline in the parent studies who were enrolled in Study GS-US-352-1154 were evaluable for splenic response assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (CCL09101/ CCL09101E/ GS-US-352-1154) | Cohort 2 (YM387-II-02/GS-US-352-1154) | Cohort 4 (GS-US-352-1672/GS-US-352-1154) | Total
Number analyzed (Participants) | 25 | 21 | 17 | 63
Participants | 20 | 19 | 6 | 45

3. Secondary Outcome: Duration of Splenic Response
Description: The interval from the first onset of splenic response (in the parent study or Study GS-US-352-1154) to the earliest date of loss of splenic response. Loss of response was defined as the reduction of splenomegaly by < 50% among responders (with splenomegaly ≥ 10 cm below the LCM at baseline) that lasts ≥ 56 days, or the recurrence of > 0 cm splenomegaly among responders (with splenomegaly > 5 and < 10 cm at baseline) that lasts ≥ 56 days.
  Duration of splenic response was measured by descriptive statistics. Data from responders who maintained their response was censored at the last assessment date.
Time Frame: as for outcome 2
Population: Duration of splenic response was assessed for spleen responders who enrolled in Study GS-US-352-1154 only.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Cohort 1 (CCL09101/ CCL09101E/ GS-US-352-1154) | Cohort 2 (YM387-II-02/GS-US-352-1154) | Cohort 4 (GS-US-352-1672/GS-US-352-1154) | Total
Number analyzed (Participants) | 20 | 19 | 6 | 45
days | 1704.5 [1153.5 to 2682.0] | 736.0 [197.0 to 1070.0] | 447.5 [128.0 to 758.0] | 990.0 [226.0 to 1802.0]

4. Secondary Outcome: Transfusion Independence Response Rate
Description: The number of transfusion dependent subjects at entry to a parent study who became transfusion-independent for ≥ 12 weeks at any time from the first dose of momelotinib in the parent study until the end of Study GS-US-352-1154.
Time Frame: From baseline in the parent study until the last assessment in Study GS-US-352-1154, up to 30 days following permanent discontinuation of momelotinib.
Population: Subjects who were transfusion dependent at baseline in the parent studies and were enrolled in Study GS-US-352-1154 were evaluable for transfusion independence response.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (CCL09101/ CCL09101E/ GS-US-352-1154) | Cohort 2 (YM387-II-02/GS-US-352-1154) | Cohort 4 (GS-US-352-1672/GS-US-352-1154) | Total
Number analyzed (Participants) | 7 | 7 | 22 | 36
Participants | 7 | 5 | 16 | 28

5. Secondary Outcome: Duration of Transfusion Independence Response
Description: The interval from the first onset date of transfusion independence (in the parent study or Study GS-US-352-1154) to the earliest date of loss of response for participants who are transfusion dependent at baseline in the parent study. Loss of TI response was defined as receiving an RBC transfusion after achieving a TI response.
  Duration of transfusion independence response was measured by descriptive statistics. Data from responders who maintained their response was censored at the last assessment date.
Time Frame: From baseline in the parent study until the last assessment date in Study GS-US-352-1154, up to 30 days following permanent discontinuation of momelotinib.
Population: Duration of transfusion independence response was assessed for transfusion independence responders who were enrolled in Study GS-US-352-1154.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Cohort 1 (CCL09101/ CCL09101E/ GS-US-352-1154) | Cohort 2 (YM387-II-02/GS-US-352-1154) | Cohort 4 (GS-US-352-1672/GS-US-352-1154) | Total
Number analyzed (Participants) | 7 | 5 | 16 | 28
days | 357.0 [117.0 to 1841.0] | 114.0 [95.0 to 126.0] | 281.5 [110.0 to 633.5] | 193.5 [110.0 to 701.0]

6. Secondary Outcome: Anemia Response Rate
Description: The number of subjects achieving an anemia response, defined as:
  * Achieving transfusion independence for ≥ 12 weeks, for subjects who were transfusion-dependent at baseline in the parent study, or
  * Having ≥ 2 g/dL increase in Hgb from baseline for ≥ 12 weeks, for subjects with Hgb < 10 g/dL at baseline in the parent study who were not transfusion-dependent (Cohort 1) or who were transfusion-independent (Cohort 2).
Time Frame: as for outcome 4
Population: Subjects who were anemia response-evaluable at baseline in the parent studies and were enrolled in Study GS-US-352-1154 were evaluable for anemia response.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (CCL09101/ CCL09101E/ GS-US-352-1154) | Cohort 2 (YM387-II-02/GS-US-352-1154) | Cohort 4 (GS-US-352-1672/GS-US-352-1154) | Total
Number analyzed (Participants) | 18 | 12 | 22 | 52
Participants | 13 | 6 | 16 | 35

7. Secondary Outcome: Duration of Anemia Response
Description: The interval from the first onset of anemia response (in the parent study or Study GS-US-352-1154) to the earliest date of loss of anemia response. Loss of anemia response was defined as having any RBC transfusion after achieving an anemia response.
  Duration of anemia response was measured by descriptive statistics. Data from responders who maintained their response was censored at the last assessment date.
Time Frame: as for outcome 4
Population: Duration of anemia response was assessed for anemia responders who were enrolled in Study GS-US-352-1154.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Cohort 1 (CCL09101/ CCL09101E/ GS-US-352-1154) | Cohort 2 (YM387-II-02/GS-US-352-1154) | Cohort 4 (GS-US-352-1672/GS-US-352-1154) | Total
Number analyzed (Participants) | 13 | 6 | 16 | 35
days | 995.0 [297.0 to 1841.0] | 120.0 [95.0 to 744.0] | 281.5 [110.0 to 633.5] | 358.0 [114.0 to 954.0]

8. Secondary Outcome: Rate of RBC Transfusion
Description: The average number of RBC units per subject month during the parent study and/or Study GS-US-352-1154.
Time Frame: From the first dose of momelotinib in the parent study until the last dose of momelotinib in Study GS-US-352-1154.
Population: as for outcome 1
Measure: Median (Full Range); unit: RBC units per month
Arm/Group | Total
Number analyzed (Participants) | 74
RBC units per month
  RBC Transfusion Rate in Parent Studies | 0.08 [0.0 to 5.4]
  RBC Transfusion Rate in Study GS-US-352-1154 | 0.00 [0.0 to 4.8]
  RBC Transfusion Rate Since 1st Dose in ParentStudy | 0.06 [0.0 to 4.9]

9. Secondary Outcome: Overall Survival
Description: The interval from the first dose of momelotinib in the parent study until death from any cause.
  Overall survival was analyzed using the Kaplan-Meier method. Data from subjects who were lost to follow-up or remained alive until the end of the study were censored at the date of last contact or last response assessment.
Time Frame: From baseline in the parent study until the date of last contact or last response assessment, up to 30 days following permanent discontinuation of momelotinib.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1 (CCL09101/ CCL09101E/ GS-US-352-1154) | Cohort 2 (YM387-II-02/GS-US-352-1154) | Cohort 4 (GS-US-352-1672/GS-US-352-1154) | Total
Number analyzed (Participants) | 30 | 22 | 22 | 74
months | NA [36.7 to 99.6] — Median not reached, reporting full range of observed values | NA [28.1 to 81.6] — Median not reached, reporting full range of observed values | NA [6.3 to 29.6] — Median not reached, reporting full range of observed values | NA [6.3 to 99.6] — Median not reached, reporting full range of observed values

10. Secondary Outcome: Progression-Free Survival
Description: The interval from the first dose of momelotinib in the parent study until the first documentation of definitive progressive disease as defined in 2006 IWG-MRT or death due to any cause.
  Subjects who were free of progression were censored at the last assessment date.
Time Frame: From baseline in the parent study until the last response assessment, up to 30 days following permanent discontinuation of momelotinib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 (CCL09101/ CCL09101E/ GS-US-352-1154) | Cohort 2 (YM387-II-02/GS-US-352-1154) | Cohort 4 (GS-US-352-1672/GS-US-352-1154) | Total
Number analyzed (Participants) | 30 | 22 | 22 | 74
months | NA [NA to NA] — Median could not be determined due to high level of censoring | NA [NA to NA] — Median could not be determined due to high level of censoring | NA [NA to NA] — Median could not be determined due to high level of censoring | NA [NA to NA] — Median could not be determined due to high level of censoring

11. Secondary Outcome: Leukemia-Free Survival
Description: The interval from the first dose of momelotinib in the parent study until the first documented leukemic transformation or death from any cause. Leukemic transformation was documented in the adverse event electronic case report form.
  Leukemia-free survival was analyzed using the Kaplan-Meier method. Subjects who were free of leukemia transformation were censored at the last assessment date.
Time Frame: From baseline in the parent study until the date of the last assessment, up to 30 days following permanent discontinuation of momelotinib.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1 (CCL09101/ CCL09101E/ GS-US-352-1154) | Cohort 2 (YM387-II-02/GS-US-352-1154) | Cohort 4 (GS-US-352-1672/GS-US-352-1154) | Total
Number analyzed (Participants) | 30 | 22 | 22 | 74
months | NA [36.7 to 99.6] — Median not reached, reporting full range of observed values | NA [28.1 to 81.6] — Median not reached, reporting full range of observed values | NA [6.1 to 29.6] — Median not reached, reporting full range of observed values | NA [6.1 to 99.6] — Median not reached, reporting full range of observed values

ADVERSE EVENTS:
Time Frame: From the first dose of momelotinib in the parent study until 30 days after the last dose in Study GS-US-352-1154.
Description: Treatment-emergent AEs were defined as AEs with onset dates on or after the start of study drug in the parent study and no later than 30 days after permanent discontinuation of study drug, or any AEs leading to premature discontinuation of study drug. It was pre-specified that adverse event data would be analyzed and summarized by starting dose in Study GS-US-352-1154. Therefore adverse event data are presented for the total subjects enrolled to Study GS-US-352-1154 and not by cohort.
Arm/Group | Total
All-Cause Mortality (participants affected / at risk) | 8/74
Serious Adverse Events (participants affected / at risk) | 49/74
Other Adverse Events (participants affected / at risk) | 73/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total (N=74)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Angina pectoris (Cardiac disorders) | 2
Aortic valve disease (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Atrioventricular block (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 4
Cardiomyopathy (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 1
Sinus node dysfunction (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 6
Ascites (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Salivary gland enlargement (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2
Varices oesophageal (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Chest pain (General disorders) | 1
Death (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 2
Cholecystitis chronic (Hepatobiliary disorders) | 1
Appendicitis (Infections and infestations) | 2
Bacterial infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis escherichia coli (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 4
Peritonitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumococcal sepsis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 7
Pneumonia klebsiella (Infections and infestations) | 1
Pneumonia pneumococcal (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Respiratory syncytial virus infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 3
Sinusitis bacterial (Infections and infestations) | 1
Systemic mycosis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Craniocerebral injury (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Tendon injury (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Intracranial venous sinus thrombosis (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient global amnesia (Nervous system disorders) | 1
Wernicke's encephalopathy (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 5
Haematuria (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total (N=74)
Anaemia (Blood and lymphatic system disorders) | 27
Leukocytosis (Blood and lymphatic system disorders) | 7
Leukopenia (Blood and lymphatic system disorders) | 9
Neutropenia (Blood and lymphatic system disorders) | 17
Thrombocytopenia (Blood and lymphatic system disorders) | 28
Thrombocytosis (Blood and lymphatic system disorders) | 4
Atrial fibrillation (Cardiac disorders) | 4
Pericardial effusion (Cardiac disorders) | 4
Sinus bradycardia (Cardiac disorders) | 7
Ear discomfort (Ear and labyrinth disorders) | 4
Cataract (Eye disorders) | 9
Dry eye (Eye disorders) | 8
Lacrimation increased (Eye disorders) | 4
Vision blurred (Eye disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 23
Abdominal pain upper (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 19
Diarrhoea (Gastrointestinal disorders) | 41
Dyspepsia (Gastrointestinal disorders) | 8
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 33
Vomiting (Gastrointestinal disorders) | 21
Asthenia (General disorders) | 5
Chest pain (General disorders) | 7
Chills (General disorders) | 4
Fatigue (General disorders) | 35
Influenza like illness (General disorders) | 4
Oedema peripheral (General disorders) | 19
Pain (General disorders) | 6
Pyrexia (General disorders) | 16
Bronchitis (Infections and infestations) | 7
Herpes zoster (Infections and infestations) | 4
Influenza (Infections and infestations) | 8
Lung infection (Infections and infestations) | 6
Sinusitis (Infections and infestations) | 14
Upper respiratory tract infection (Infections and infestations) | 14
Urinary tract infection (Infections and infestations) | 23
Contusion (Injury, poisoning and procedural complications) | 22
Fall (Injury, poisoning and procedural complications) | 8
Foot fracture (Injury, poisoning and procedural complications) | 4
Activated partial thromboplastin time prolonged (Investigations) | 5
Alanine aminotransferase increased (Investigations) | 19
Amylase increased (Investigations) | 12
Aspartate aminotransferase increased (Investigations) | 11
Blood alkaline phosphatase increased (Investigations) | 5
Blood bilirubin increased (Investigations) | 8
Blood creatinine increased (Investigations) | 17
Blood uric acid increased (Investigations) | 4
Electrocardiogram QT prolonged (Investigations) | 4
Gamma-glutamyltransferase increased (Investigations) | 4
International normalised ratio increased (Investigations) | 5
Lipase increased (Investigations) | 15
Lymphocyte count decreased (Investigations) | 4
Neutrophil count decreased (Investigations) | 5
Platelet count decreased (Investigations) | 11
Weight decreased (Investigations) | 8
Weight increased (Investigations) | 4
White blood cell count decreased (Investigations) | 5
Decreased appetite (Metabolism and nutrition disorders) | 10
Dehydration (Metabolism and nutrition disorders) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 11
Hyperuricaemia (Metabolism and nutrition disorders) | 18
Hypocalcaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 21
Back pain (Musculoskeletal and connective tissue disorders) | 12
Bone pain (Musculoskeletal and connective tissue disorders) | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18
Dizziness (Nervous system disorders) | 28
Dysgeusia (Nervous system disorders) | 5
Headache (Nervous system disorders) | 28
Hypoaesthesia (Nervous system disorders) | 5
Neuropathy peripheral (Nervous system disorders) | 19
Paraesthesia (Nervous system disorders) | 5
Peripheral sensory neuropathy (Nervous system disorders) | 31
Syncope (Nervous system disorders) | 4
Anxiety (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 7
Insomnia (Psychiatric disorders) | 13
Acute kidney injury (Renal and urinary disorders) | 5
Pollakiuria (Renal and urinary disorders) | 6
Proteinuria (Renal and urinary disorders) | 5
Urinary retention (Renal and urinary disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 8
Night sweats (Skin and subcutaneous tissue disorders) | 10
Petechiae (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 10
Rash (Skin and subcutaneous tissue disorders) | 12
Skin lesion (Skin and subcutaneous tissue disorders) | 4
Skin ulcer (Skin and subcutaneous tissue disorders) | 4
Tooth extraction (Surgical and medical procedures) | 5
Flushing (Vascular disorders) | 8
Haematoma (Vascular disorders) | 5
Hypertension (Vascular disorders) | 14
Hypotension (Vascular disorders) | 16

LIMITATIONS AND CAVEATS:
Cohort 3 was discontinued and excluded from the safety and efficacy analyses.

The survival analyses were subject to a high level of censoring.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Most restrictive: Site may not present or publish results of Trial without advance written notice of Sponsor or two years after completion of Trial at all participating sites. Site must submit all proposed publications or presentations to Sponsor for review. Sponsor can review communications prior to public release and embargo trial results communications for a period between 75 and 180 days from submission to Sponsor for review. Sponsor has right to request Site remove Confidential Information.

DOCUMENTS (2):
  • Study Protocol (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT02124746/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/46/NCT02124746/SAP_001.pdf